CLINICAL TRIAL: NCT01199445
Title: Efficacy of Vitamin A in Fortified Extruded Rice in School Children in Satun, Thailand
Brief Title: Efficacy of Vitamin A in Fortified Extruded Rice in School Children
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Mahidol University (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ETH2010/SP02
Record Dates: First submitted 2010-08-20; First posted 2010-09-13 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2012-06

CONDITIONS: Vitamin A Deficiency
Keywords: vitamin A deficiency
MeSH Terms: conditions — Vitamin A Deficiency | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- triple fortified extruded rice (Experimental)
  Interventions: Dietary Supplement: Triple fortified extruded tice (Fe, Zn and vitamin A)
- regular meal (Other): regular vitamin A meal
  Interventions: Dietary Supplement: Triple fortified extruded tice (Fe, Zn and vitamin A)

INTERVENTIONS:
Dietary Supplement: Triple fortified extruded tice (Fe, Zn and vitamin A) — Triple fortified extruded rice (Fe, Zn and vitamin A)will be mix at ratio of 1:50 with normal rice then give to children at school lunch meal for 60 days.

SUMMARY:
The project aims to evaluate the potential impact triple fortified rice grains, mixed into natural rice grains, can have on vitamin A status if fed to school children in Southern Thailand. Within a 60 day intervention study, changes in vitamin A status in young children fed the fortified rice compared to children consuming non-fortified rice will be assessed.

DETAILED DESCRIPTION:
Iron, zinc and vitamin A deficiencies are particularly common among children and young women in developing countries of South and Southeast Asia. Rice is a common staple for a large part of these sub-regions of Asia. In spite of a wide range of rice varieties eaten, rice is eaten by all age groups and is one of the first few foods used as complementary food for infants.

Fe fortification of rice using a method of heat extrusion and micronized ferric pyrophosphate (FePP) as iron fortificant has shown to be efficacious in increasing iron stores and reducing the prevalence of iron deficiency in Indian school children. Subsequent extrusion trials have shown promising results with respect to color and vitamin A (VA) stability when rice grains were triple fortified with Fe, Zn and vitamin A.

Preliminary data in the region of Satun, South Thailand, have shown that zinc and vitamin A intakes are low. Biochemical indicators have confirmed zinc deficiency and suboptimal vitamin A status in 1/3 of school aged children. Since rice is the main staple food in this area, rice triple fortified with Fe, VA and Zn is a promising strategy to combat micronutrient deficiencies in children.

The aim of this study is to demonstrate whether triple fortified rice has an impact on vitamin A status of children. The study will be conducted in school children (8 to 12 years old). The children will be randomized to either receive a daily lunch rice meal prepared from fortified rice (the triple fortified rice grains will be mixed into natural rice at a ratio of 1:50) or from non-fortified rice for 60 days. As serum retinol concentration, the most widely used indicator for the assessment of vitamin A status, is not a very reliable indicator due to homeostatic control and the influence of infection, we will in addition use the tracer methodology using dilution of stable isotopes with which total body vitamin A pool size will be estimated prior to the intervention and after 60 days of the intervention..

ELIGIBILITY:
Inclusion Criteria:

* Children, aged 8-12 years, both sexes, attending the local primary schools
* No known or reported history of significant chronic illness
* Free of acute illness and febrile and gastrointestinal problems

Exclusion Criteria:

* Children with severe vitamin A deficiency with a clinical sign of Bioit's spot or ocular signs of xerophthalmia will be excluded
* Children who have serum retinol < 0.7 umol/L

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Vitamin A in the entire body | 4 months
  A quantitative estimate of the size of exchangeable body pool of vitamin A. The exchangeable body pool of vitamin A refer to the vitamin A in body that is in dynamic state.

SECONDARY OUTCOMES:
Serum retinol | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Hurrell, Ph.D, Principal Investigator — Swiss Federal Institute of Technology (ETH,Zurich)
Locations (1):
- Tessaban 3 School, Muang, Changwat Satun, Thailand

REFERENCES:
- [Derived] Pinkaew S, Wegmuller R, Wasantwisut E, Winichagoon P, Hurrell RF, Tanumihardjo SA. Triple-fortified rice containing vitamin A reduced marginal vitamin A deficiency and increased vitamin A liver stores in school-aged Thai children. J Nutr. 2014 Apr;144(4):519-24. doi: 10.3945/jn.113.182998. Epub 2014 Feb 5. PMID 24500930